CLINICAL TRIAL: NCT05236907
Title: The Efficacy of Oral Melatonin in Preventing Postoperative Delirium for Patients Undergoing Orthopedic Surgery Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Melatonin123
Record Dates: First submitted 2022-01-06; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Delirium, Anesthesia Emergence; Delirium
Keywords: Delirium; melatonin; patients; surgery; postoperative; benzodiazepines; orthopedic; preoperatively
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Melatonin; Midazolam

STUDY DESIGN:
Intervention Model Description: Patients were divided into three groups at random, with 12 patients in each group, using a double-blinded method.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It has been done on all the study's contributors and workers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Placebo Comparator): Patients in this group received nothing for sedation.
  Interventions: Other: No intervention
- Midazolam group (Active Comparator): 7.5 mg of Midazolam were given orally the night before operation. Another dose 90 min. preoperatively.
  Interventions: Drug: Midazolam
- Melatonin group (Experimental): 5 mg of Melatonin were given orally the night before operation. Another dose 90 min. preoperatively
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — The patients were assessed using the Memorial Delirium Assessment Scale (MDAS) after the operation at 30, 60, and 90 min. Melatonin was shown to reduce delirium from 41.6% to 16.6% at 60 minutes, and the significant reduction was at 90 minutes (0%) when compared to both groups. Thus, melatonin was found to be successful in decreasing postoperative delirium when administered preoperatively.
  Other Names: Midazolam
  Arms: Melatonin group
Other: No intervention — No intervention was used.
  Arms: Control Group
Drug: Midazolam — 7.5 mg of Midazolam orally.
  Arms: Midazolam group

SUMMARY:
Postoperative delirium is a complication that should not be underestimated. As it elaborates many complications that could be avoided when an accurate assessment of the risk factors and interventional measures are taken appropriately when needed.

DETAILED DESCRIPTION:
Delirium is a variation in concentration capabilities that occurs acutely in association with a disturbed level of consciousness. Delirium is more common in orthopaedic surgery patients than in general surgery patients. As delirium ratios range from 44% to 55% in hip surgery patients, otherwise only 10%-14% of general surgery patients. Several studies were carried out and found that melatonin levels correlate with the development of delirium postoperatively. This study was conducted to determine the efficacy of administering melatonin preoperatively in patients undergoing orthopedic surgery to prevent postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

1- Patients in good general health. 2. Baseline MDAS <13. 3. No seizure disorder.

Exclusion Criteria:

1. Patients with a neurological disorder (e.g., dementia, stroke, epilepsy).
2. Patients with a history of acute or chronic confusion.
3. Patients taking centrally acting drugs (e.g., antidepressants, antiparkinsonian drugs, sedatives, monoamine oxidase inhibitors), or alcohol abusers.
4. Patients who have medical disorders predisposing to delirium (e.g. cachexia, thyroid dysfunction, renal failure).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of oral Melatonin in preventing Postoperative Delirium after general anesthesia | 1 week
  This interventional trial is done to determine the efficacy of preoperative melatonin administration in reducing postoperative delirium rates.

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - Al-Kadhemya Private Hospital, Baghdad
  - Ghazi Al-Hariri Teaching Hospital, Baghdad

IPD SHARING:
Plan to Share IPD: No